CLINICAL TRIAL: NCT02150291
Title: A Pilot Study to Assess the Efficacy and Safety of Folic Acid and/or Vitamin B Complex on Hepatitis C Infected Patients Treated With Pegylated Interferon and Ribavirin.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: British University In Egypt (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nermeen Nabil Ashoush, Lecturer Assistant in Clinical Pharmacy Department, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2107
Record Dates: First submitted 2014-05-27; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Folic Acid; Vitamin B Complex

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Active Comparator): one capsule of 5 mg of Folic acid twice daily and a tablet of Neurobion three times per day during hepatitis C treatment
  Interventions: Dietary Supplement: Folic acid; Drug: Neurobion
- Group B (Active Comparator): Patients will receive one capsule of 5 mg of Folic acid twice daily during hepatitis C treatment
  Interventions: Dietary Supplement: Folic acid
- Group C (Active Comparator): Patients will receive a tablet of Neurobion three times per day during hepatitis C treatment
  Interventions: Drug: Neurobion
- Group D (Placebo Comparator): Patients will receive matching placebo capsule to take during hepatitis C treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Dietary Supplement: Folic acid
  Arms: Group A; Group B
Drug: Neurobion
  Arms: Group A; Group C
Drug: placebo
  Arms: Group D

SUMMARY:
Since success of the combination therapy with PEG-IFN and RBV is contingent on maintaining adequate doses of both drugs throughout the treatment period, the emergence of hematological side effects is expected and requires intervention. The hematological adverse effects lead to a trade-off between continuing the treatment with optimal dosage, to clear the virus, exacerbating thereby the side effects versus decreasing dosage to relieve severe anemia, reducing thereby the chances of achieving sustained virological response (SVR). Therefore, we aimed at giving Folic acid® and Neurobion® to HCV-infected patients during treatment with different types of PEG-IFN plus ribavirin in an attempt to evaluate its efficacy and safety as a prophylactic treatment to prevent hematological adverse effects. Preventing adverse effects without interfering with the therapeutic efficacy of different types of PEG-IFN plus ribavirin in HCV patients will lead to better health outcomes and improvement in their quality of life (HRQOL).

ELIGIBILITY:
Inclusion Criteria:

Chronic hepatitis C patients of both sexes were eligible for inclusion if they were HCV RNA positive, naive to PEG-INF and RBV, and had abnormal serum alanine transaminase levels on two occasions during the preceding six months.

Exclusion Criteria:

Patients with significant hematological abnormalities at baseline, such as neutropenia (ANC <1200 x 103 cells/µL), thrombocytopenia (<70 x 103 cells/ µL), and anemia (<10.5 g/dL), were excluded. Patients were also excluded from study participation if they had serum creatinine ≥1.70 mg/dL (150 µmol), hepatitis B surface antigen positivity, decompensated cirrhosis, or other forms of liver disease not attributable to HCV. Patients with severe depression or psychosis, uncontrolled seizures, poorly controlled cardiovascular disease, diabetes mellitus, or autoimmune disorders were also ineligible. Women were ineligible for study participation if they were pregnant or unwilling to use at least 2 forms of effective contraception during the entire study period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Effect of folic acid and/or Vitamin B complex to prevent adverse effect of pegylated interferon and ribavirin | 1 YEAR
  Maintain absolute neutrophil count (ANC) levels >750 cells/mm3, hemoglobin levels >10.5 g/dL to prevent adjustment to the PEG-INF dose or its temporary suspension. Moreover, to maintain a sustained platelet level above 45,000 platelet/mm3. During therapy thrombocytopenia was assessed at levels of 50,000 and 25,000/µl, since these levels are the usual thresholds for dose reductions or discontinuation of peginterferon alfa/ribavirin therapy.

SECONDARY OUTCOMES:
Effect of folic acid and/or Vitamin B complex on the efficacy of pegylated interferon and ribavirin. | 1 year and 6 month after end of treatment
  Biochemical improvement of liver function and sustained virological response (SVR). Biochemical improvement was defined as a decrease in alanine transaminase (ALT) level and Aspartate transaminase (AST). A sustained virological response (SVR) is deﬁned as undetectable serum HCV RNA (< 51 IU/ml) 24 weeks after the completion of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Abbasiya, Egypt